CLINICAL TRIAL: NCT03485313
Title: Clinical Evaluation to Determine the Expected Values Distribution of β-hCG for the RAMP® Total β-hCG Test in a Healthy, Non-pregnant Reference Population
Brief Title: Beta-hCG Test Reference Range Determination
Status: Terminated | Type: Observational
Why Stopped: Study stopped due to slow enrollment; sufficient data collected for analysis.
Sponsor: Response Biomedical Corp. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP027
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Healthy
Keywords: Healthy; Volunteer; Female; Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA blood samples will be processed into plasma and stored frozen for study duration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, single-centre study to determine the reference range (95th percentile) of human chorionic gonadotropin (hCG) levels in a healthy, non-pregnant, adult female population using the RAMP® Total β-hCG test.

DETAILED DESCRIPTION:
Human chorionic gonadotropin (hCG) is a glycoprotein hormone secreted by the placenta shortly after implantation of a fertilized ovum into the uterine wall and the rapid rise of blood hCG concentration after conception makes it an excellent marker for confirmation and monitoring of early pregnancy. As such, levels in the blood of non-pregnant premenopausal individuals are low, typically < 5 mIU/mL (milli-International Unit per milliliter).

In terms of identifying a clinically significant range of expected hCG values as determined by the RAMP β-hCG test, a 95th percentile of a healthy, non-pregnant, adult female reference population [upper reference limit (URL)] shall be determined in this study.

Subjects who meet the inclusion and exclusion criteria, and give informed consent will be enrolled in this study. Because hCG levels in blood increase with age, the study population will be divided into two age groups: 18 to 40 years and >40 years, with approximately 125 subjects per group.

One EDTA (ethylenediaminetetraacetic acid) blood sample will be collected from each subject via standard venipuncture. The maximum trial duration for each subject will be one visit/blood draw.

ELIGIBILITY:
Inclusion Criteria:

1. Apparently healthy, non-pregnant females, of any race.
2. >18 years of age.
3. Willing to voluntarily agree to sign a consent form.

Exclusion Criteria:

1. Current pregnancy, suspected pregnancy, or pregnancy within previous 12 months.
2. Currently lactating/nursing a child.
3. Current diagnosis of Gestational Trophoblastic Disease, Gestational Trophoblastic Tumor or Gestational Trophoblastic Neoplasia.
4. Current diagnosis of non-trophoblastic tumors.
5. Current diagnosis of cancer and/or has undergone immunotherapy in the previous 12 months.
6. Current diagnosis of a serious health condition that involves inpatient care or continuing treatment by a health care provider, such as:

   * Conditions or treatments that result in continuous or episodic incapacity (e.g. pneumonia, epilepsy).
   * Permanent or long-term conditions (e.g. HIV, Alzheimer's, severe stroke).
   * Conditions requiring multiple treatment/recovery cycles (e.g. kidney disease).
7. Hospitalization (for >24 hours) or major surgery within previous 3 months.
8. Unable, or unwilling, to provide required blood sample for testing.
9. Investigator believes subject is unsuitable for inclusion in the trial (i.e. has serious condition(s) or other reason(s) that could limit their ability to participate in the study; or impact the scientific integrity of the study).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately two hundred-fifty (250) healthy, non-pregnant adult female subjects will be enrolled in the study. Because hCG levels in blood increase with age, the study population will be divided into two age groups: 18 to 40 years and >40 years, with approximately 125 subjects per group.There are no enrollment restrictions based upon race or ethnic origin.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
Measurement of blood hCG level. | baseline
  Measurement of hCG in a single EDTA blood sample from healthy, non-pregnant adult female subjects using the RAMP Total β-hCG test.

CONTACTS AND LOCATIONS:
Locations (1):
- Response Biomedical Corp., Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No